CLINICAL TRIAL: NCT03084757
Title: SHIVA02 - Evaluation of the Efficacy of Targeted Therapy Based on Tumor Molecular Profiling in Patients With Advanced Cancer Using Each Patient as Its Own Control
Brief Title: SHIVA02 - Evaluation of the Efficacy of Targeted Therapy Based on Tumor Molecular Profiling in Patients With Advanced Cancer Using Each Patient as Its Own Control (SHIVA02)
Acronym: SHIVA02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IC 2016-06
Record Dates: First submitted 2017-03-02; First posted 2017-03-21 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Cancer; Solid Tumor, Adult
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- research of druggable molecular alterations on tumor biopsy (Experimental)
  Interventions: Diagnostic Test: research of druggable molecular alterations on tumor biopsy

INTERVENTIONS:
Diagnostic Test: research of druggable molecular alterations on tumor biopsy — The study will run in 2 steps. Before starting a new treatment, patients with advanced cancer will undergo a tumor biopsy of a metastatic site in order to perform molecular analyses seeking for druggable molecular alterations

SUMMARY:
The study will evaluate the efficacy of targeted therapy based on tumor molecular profiling versus conventional chemotherapy in patients with advanced cancer using each patient as its own control. This study is a study involving patients with advanced cancer. All types of solid tumors will be allowed in the study.

ELIGIBILITY:
Inclusion criteria:

Inclusion will proceed in 2 steps. First step for molecular analyses and second step in order to be included in the efficacy analysis.

Inclusion criteria for Step 1:

1. Patient with recurrent/metastatic solid tumor who failed or are not candidate for treatments usually proposed in first intention and for whom a prospective clinical trial has been indicated in a tumor board
2. Patient with a documented progression before the start of conventional therapy according to RECIST 1.1.
3. Patient ≥18 years old

3) Disease amenable to biopsy 5) ECOG performance status of 0 or 1 6) Measurable disease 7) Adequate renal function defined by a serum creatinine <1.5xUNL (upper normal limit) 8) Adequate liver function test defined by SGOT & SGPT <3xUNL (5xUNL in case of liver metastases), and bilirubin level <1.5xUNL 9) Adequate bone marrow function defined by platelets >100,000/mm3, hemoglobin >9 g/dL, and neutrophils >1,000/mm3 10) Patient must be affiliated to the French Social Security System 11) Signed informed consent 12 For female of child-bearing potential: a negative pregnancy test <72 hours before starting study treatment is required. If sexually active, female of childbearing potential must use "highly effective" methods of contraception for the study duration and for 3 months following the last treatment 13) For male of reproductive potential: any sexually active male patient must use a condom while on study treatment and for 3 months following the last treatment

Inclusion criteria for Step 2:

1. Patient for whom the Molecular Biology Board (MBB) has identified a druggable molecular alteration of the RAF/MEK signaling pathway and a treatment recommendation has been established by the MBB.
2. Patient with a documented progression during the conventional therapy according to RECIST 1.1.
3. Patient with imaging performed within 28 days prior to the planned start date of treatment

Exclusion criteria:

1. Patients below 18 years old
2. Patients with CNS involvement that has not been controlled for >3 months
3. Patients planned to receive a molecularly targeted agent
4. Patients who are candidate to receive a molecularly targeted agent that is approved for their disease
5. Patients with other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study, including uncontrolled diabetes, cardiac disease, uncontrolled hypertension, congestive cardiac failure, ventricular arrhythmias, active ischemic heart disease, myocardial infection within one year, chronic liver or renal disease, active gastrointestinal tract ulceration, severely impaired lung function
6. Pregnant and/or breastfeeding women
7. Patients individually deprived of liberty or placed under the authority of a tutor
8. Patients with any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
9. Known HIV, HBV, or HCV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a PFS2 to PFS1 ratio superior to 1.5. | 3 years
  PFS1 is defined as the time to a documented progression under conventional therapy according to RECIST 1.1. PFS2 is defined as the time to a documented progression or death when patients are treated by targeted therapy according to RECIST 1.1

SECONDARY OUTCOMES:
Overall response rate (ORR) on both treatments | 3 years
  Evaluation of the best objective response rate (ORR) for each treatment according to RECIST 1.1 The best ORR is the best response reached during treatment according to RECIST 1.1 criteria.
Overall survival (OS) | 3 years
  Evaluation of overall survival (OS) defined as the time between inclusion and death, whatever the cause is. Alive patients will be censored at their last known contact date.
number of grade 3 or 4 adverse events and grade 1 or 2 adverse events that lead to dose modification or interruption | 3 years
  Evaluation of toxicities related to treatments according to CTCAE v4.03. Only grade 3 or 4 adverse events and grade 1 or 2 adverse events that lead to dose modification or interruption
Ability of ctDNA to detect molecular alterations identified on tumor biopsies | at baseline
  Percentage of patients for whom all druggable molecular alterations detected on the tumor biopsy are also detected on ctDNA.
Ability of fine-needle aspiration cytology to detect molecular alterations identified on tumor biopsies | at baseline
  Percentage of patients for whom all druggable molecular alterations detected on the tumor biopsy are also detected on fine-needle aspiration cytology
Ability of sequential ctDNA sampling to predict response/resistance to treatment | through study completion, every 2 months
  Changes in ctDNA levels and molecular alterations observed at different time points.
Proportion of patients with a PFS2 to PFS1 ratio superior to 1.5, including patients who were treated with matched therapy based on a molecular alteration outside of RAF/MEK pathway | 3 years
  PFS1 is defined as the time to a documented progression under conventional therapy according to RECIST 1.1. PFS2 is defined as the time to a documented progression or death when patients are treated by targeted therapy according to RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Institut Bergonié, Bordeaux
  - Centre LEON BERARD, Lyon
  - Institut Curie, Paris
  - Institut Curie Hôpital René Huguenin, Saint-Cloud

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share de-identified data sets with interested researchers, educators or clinicians. Materials generated under the project will be disseminated in accordance with Institut Curie policies.
Time Frame: Data requests can be submitted starting 9 months after article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific reserach, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).

REFERENCES:
- [Derived] Dupain C, Masliah-Planchon J, Gu C, Girard E, Gestraud P, Du Rusquec P, Borcoman E, Bello D, Ricci F, Hescot S, Sablin MP, Tresca P, de Moura A, Loirat D, Frelaut M, Vincent-Salomon A, Lecerf C, Callens C, Antonio S, Franck C, Mariani O, Bieche I, Kamal M, Le Tourneau C, Servois V. Fine-needle aspiration as an alternative to core needle biopsy for tumour molecular profiling in precision oncology: prospective comparative study of next-generation sequencing in cancer patients included in the SHIVA02 trial. Mol Oncol. 2021 Jan;15(1):104-115. doi: 10.1002/1878-0261.12776. Epub 2020 Sep 15. PMID 32750212